CLINICAL TRIAL: NCT06535230
Title: Does Induction of Anesthesia with Target-controlled Propofol Infusion Reduce the Risk of Post-induction Hypotension in High-risk Patients?
Brief Title: Anesthesia Induction with the Target-controlled Infusion of Propofol in High-risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ATADEK-2024
Record Dates: First submitted 2024-07-18; First posted 2024-08-02 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia; Hemodynamic Instability
Keywords: Anesthesia induction; Post-induction hypotension; Target controlled infusions; High-risk patients
MeSH Terms: interventions — Hemodynamic Monitoring

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, non-blinded, randomized controlled trial. Patients were allocated to 2 groups:
  Group 1: Patients who underwent manual anesthesia induction Group 2 : Patients who underwent anesthesia induction with target-controlled infusion,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who were assigned to have manual anesthesia induction group with propofol (Active Comparator): Patients who were assigned to have a manual anesthesia induction group, propofol was administered 1-2 mg/kg in 1-2 minutes to achieve a level of hypnosis measured by bispectral index ( BIS ) of 35-60
  Interventions: Drug: Manual anesthesia induction; Device: Hemodynamic monitoring with pressure recording analytical method (PRAM)
- Patients who were assigned to have target controlled infusions ( TCI) induction with propofol (Active Comparator): Patients who were assigned to have TCI induction had the target effect site concentration (Ce) of propofol (Ce) set at 1 μg ml-1 using the Schneider model and subsequently modified to achieve and maintain a level of hypnosis measured by BIS of 35-55
  Interventions: Drug: Anesthesia induction with Target controlled infusions (TCI); Device: Hemodynamic monitoring with pressure recording analytical method (PRAM)

INTERVENTIONS:
Drug: Manual anesthesia induction — In manual anesthesia induction, anesthetic agents are administered at a fixed dose and rate adjusted according to the patient's weight
  Other Names: Manuel induction
  Arms: Patients who were assigned to have manual anesthesia induction group with propofol
Drug: Anesthesia induction with Target controlled infusions (TCI) — Target controlled infusion (TCI) system aims to reach the theoretically targeted blood or brain concentration of anesthetic agents based on the patient's age, weight, and height, with computer-assisted algorithms.
  Other Names: TCI induction
  Arms: Patients who were assigned to have target controlled infusions ( TCI) induction with propofol
Device: Hemodynamic monitoring with pressure recording analytical method (PRAM) — The pulse contour device MostCare (Vytech, Vygon, Padova, Italy) provides functional hemodynamic monitoring using the pressure recording analytical method.

SUMMARY:
The purpose of this study is to compare the risk of hypotension following induction of anesthesia in high-risk patients (American Society of Anesthesiologists risk scores III and IV) using target-controlled infusion (TCI) of propofol versus standard manual induction of anesthesia. Our previously published study compared TCI and manual induction of anesthesia in a general patient population and found that hypotension developed less with TCI induction. This study is a continuation of the other study and will be conducted in high-risk patients.

DETAILED DESCRIPTION:
Hypotension after induction of anesthesia is a very common condition. Despite well-known risk factors and advanced monitoring techniques, hypotension after induction of anesthesia occurs in approximately 30% of patients. The risk of hypotension increases in patients with comorbidities such as hypertension, heart failure, renal failure, diabetes mellitus, patients with high ASA (American Society of Anesthesiologists ) risk scores, geriatric patients, patients undergoing major surgery, and patients with prolonged fasting periods. In order to prevent post-induction hypotension, the risk factors of the patient (such as comorbidities, and surgery) cannot be changed, but this risk can be reduced with different anesthesia induction techniques.

Since anesthetic agents are administered at a fixed dose and rate adjusted according to the patient's weight in standard anesthesia induction, it may cause hypotension in patients with low cardiovascular performance.

The fall in blood pressure is due to a decrease in systemic vascular resistance or cardiac output and may be increased by the concomitant use of other drugs such as remifentanil. Target-controlled infusions (TCI) have been developed to overcome these drawbacks of standard anesthesia induction and maintenance. TCI systems enable titration of anesthetic agents according to the needs of each patient by using pharmacokinetic models through perfusers with special microprocessors. With these features, TCI can provide better control of hemodynamic variations during induction and maintenance of anesthesia. Patients will undergo hemodynamic monitoring using the pressure analytic recording method (PRAM). The functional hemodynamic data provided by this monitoring technique will allow us to better analyze the causes and consequences of hypotension. In this study, investigators aimed to monitor and compare the hemodynamic effects of TCI induction and manual anesthesia induction through PRAM parameters by monitoring patients with high ASA scores before and after induction. Investigators anticipate that these 2 technologies (TCI and PRAM) can provide a better hemodynamic profile in the high-risk patient group with high ASA scores thanks to the advanced monitoring provided to the patient in our anesthesia practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the American Society of Anesthesiology physical status 3-4
* Underwent major elective surgery
* Required intra-arterial blood pressure monitoring before induction.

Exclusion Criteria:

* Under 18 years of age
* Patients with the American Society of Anesthesiology physical status 1-2
* Arrhythmia (atrial fibrillation, frequent premature beat)
* Severe valvular heart disease
* Morbid obesity
* Intubation difficulty
* Drug addiction
* Treatment with opiates
* Pregnancy
* Emergency surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic arterial pressure (SAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Systolic arterial pressure (SAP- mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SAP is a parameter used to assess the pressure of the arterial system during cardiac systole
Diastolic arterial pressure (DAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Diastolic arterial pressure (DAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). DAP is a parameter used to assess the pressure of the arterial system during cardiac diastole
Mean arterial pressure (MAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Mean arterial pressure (MAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). MAP is a parameter used to assess organ perfusion

SECONDARY OUTCOMES:
Arterial elastance (Ea) measured before anesthesia induction was investigated whether is a predictive parameter for post-induction hypotension in patients undergoing general anesthesia with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Ea ((mmHg m-2ml-1)is an indicator of cardiac afterload and arterial tone and can be calculated by the ratio of the end-systolic pressure (ESP) and stroke volume (SV) obtained from arterial wave analysis. Ea was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy) before the anesthesia induction
Stroke volume variation (SVV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI and manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Stroke volume variation (SVV,%), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SVV is a parameter used to asses cardiac preload and fluid responsiveness
Pulse pressure variation (PPV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Pulse pressure variation (PPV,%) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). PPV is a parameter used to asses cardiac preload and fluid responsiveness.
Cardiac power output (CPO), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac power output (CPO, Watt) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CPO is a parameter used to asses cardiac reserve
Cardiac index (CI), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac index (CI, L/min/m2), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CI is a parameter used to asses cardiac stroke volume
Dp/Dt, measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Dp/Dt(mmHg/msn), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). Dp/Dt is a parameter used to asses cardiac contractility
Heart rate (HR), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Heart rate (HR/bpm) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). HR is a parameter used to assess the cardiac rate.

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi Toraman, M.D., Study Director — Acibadem Mehmet Ali Aydinlar University School of Medicine, Department of Anesthesiology
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saugel B, Sessler DI. Perioperative Blood Pressure Management. Anesthesiology. 2021 Feb 1;134(2):250-261. doi: 10.1097/ALN.0000000000003610. No abstract available. PMID 33206118
- [Background] Sessler DI, Khan MZ, Maheshwari K, Liu L, Adegboye J, Saugel B, Mascha EJ. Blood Pressure Management by Anesthesia Professionals: Evaluating Clinician Skill From Electronic Medical Records. Anesth Analg. 2021 Apr 1;132(4):946-956. doi: 10.1213/ANE.0000000000005198. PMID 33031346
- [Background] Billard V, Moulla F, Bourgain JL, Megnigbeto A, Stanski DR. Hemodynamic response to induction and intubation. Propofol/fentanyl interaction. Anesthesiology. 1994 Dec;81(6):1384-93. doi: 10.1097/00000542-199412000-00013. PMID 7992907
- [Background] Gao Q, Sun L. Hypotension during induction: prediction or prevention? J Anesth. 2020 Apr;34(2):308. doi: 10.1007/s00540-019-02710-9. Epub 2019 Nov 9. No abstract available. PMID 31707517
- [Background] Kazama T, Ikeda K, Morita K, Kikura M, Doi M, Ikeda T, Kurita T, Nakajima Y. Comparison of the effect-site k(eO)s of propofol for blood pressure and EEG bispectral index in elderly and younger patients. Anesthesiology. 1999 Jun;90(6):1517-27. doi: 10.1097/00000542-199906000-00004. PMID 10360846
- [Background] Yildirim SA, Dogan L, Sarikaya ZT, Ulugol H, Gucyetmez B, Toraman F. Hypotension after Anesthesia Induction: Target-Controlled Infusion Versus Manual Anesthesia Induction of Propofol. J Clin Med. 2023 Aug 14;12(16):5280. doi: 10.3390/jcm12165280. PMID 37629322